CLINICAL TRIAL: NCT01126918
Title: Eating Disorders Prevention: An Effectiveness Trial for At-Risk College Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Collaborators: University of Texas at Austin (Other); Drexel University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MH086582
Record Dates: First submitted 2010-05-18; First posted 2010-05-20 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Eating Disorders; Obesity
Keywords: Eating Disorders; Obesity; Body Dissatisfaction; Female
MeSH Terms: conditions — Feeding and Eating Disorders; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Brochure Condition (Active Comparator): Participants in this condition receive an educational brochure about healthy body image via post-mail.
  Interventions: Behavioral: Body Project
- Group Condition (Experimental): Participants in this condition attend four 1-hour group meetings (one per week for four consecutive weeks) in which they complete a series of written and verbal exercises intended to increase body satisfaction.
  Interventions: Behavioral: Body Project

INTERVENTIONS:
Behavioral: Body Project — Participants in this intervention attend four 1-hour group meetings (one per week for four consecutive weeks) in which they complete a series of written and verbal exercises intended to increase body satisfaction.

SUMMARY:
This three-site effectiveness trial will test whether a brief dissonance-based eating disorder prevention program produces intervention effects when college counselors, psychologists, and nurses are responsible for participant recruitment, screening, and intervention delivery under ecologically valid conditions.

DETAILED DESCRIPTION:
Threshold and subthreshold eating disorders affect over 10% of young women and are associated with functional impairment, distress, psychiatric comorbidity, medical complications, mortality, and risk for obesity onset. Accordingly, a pressing public healthy priority is to develop effective prevention programs for eating pathology. The proposed project will be the first effectiveness trial to test whether an eating disorder prevention program with strong empirical support from efficacy trials produces effects under ecologically valid conditions among high-risk female college students, which is a vital step toward widespread dissemination of programs developed with NIH funding. The proposed cost-effectiveness analyses and examination of process factors that predict larger intervention effects will also represent novel contributions to the literature.

ELIGIBILITY:
Inclusion Criteria:

* (1) is a registered student at a participating school, (2) self-reports body image concerns

Exclusion Criteria:

* meets DSM-IV criteria for anorexia nervosa, bulimia nervosa, or binge eating disorder

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2010-04; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
eating disorder symptoms, risk for future eating disorder and obesity onset | 2 years

SECONDARY OUTCOMES:
mediators to intervention effects | 2 years
  We will test whether the dissonance program intervention effects are mediated by change in thin-ideal internalization
moderators to program effects | 2 years
  We will test whether certain factors moderate program effects (e.g., initial body dissatisfaction level).

CONTACTS AND LOCATIONS:
Overall Officials: Eric Stice, Ph.D., Principal Investigator — Oregon Research Institute; Meghan Butryn, Ph.D., Principal Investigator — Drexel University
Locations (7):
- United States (7):
  - Northwest Christian University, Eugene, Oregon
  - University of Oregon, Eugene, Oregon
  - Drexel University, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - University of Texas at Austin, Austin, Texas
  - Southwestern University, Georgetown, Texas

REFERENCES:
- [Derived] Stice E, Desjardins C, Shaw H, Siegel S, Gee K, Rohde P. Prevalence, incidence, impairment, course, and diagnostic progression and transition of eating disorders, overweight, and obesity in a large prospective study of high-risk young women. J Psychopathol Clin Sci. 2025 May;134(4):427-437. doi: 10.1037/abn0000965. Epub 2024 Nov 7. PMID 39509183
- [Derived] Stice E, Desjardins CD, Rohde P. Young women who develop anorexia nervosa exhibit a persistently low premorbid body weight on average: A longitudinal investigation of an important etiologic clue. J Psychopathol Clin Sci. 2022 Jul;131(5):479-492. doi: 10.1037/abn0000762. Epub 2022 Jun 2. PMID 35653756
- [Derived] Stice E, Desjardins CD, Rohde P, Shaw H. Sequencing of symptom emergence in anorexia nervosa, bulimia nervosa, binge eating disorder, and purging disorder and relations of prodromal symptoms to future onset of these disorders. J Abnorm Psychol. 2021 May;130(4):377-387. doi: 10.1037/abn0000666. PMID 34180702
- [Derived] Stice E, Rohde P, Shaw H, Desjardins C. Weight suppression increases odds for future onset of anorexia nervosa, bulimia nervosa, and purging disorder, but not binge eating disorder. Am J Clin Nutr. 2020 Oct 1;112(4):941-947. doi: 10.1093/ajcn/nqaa146. PMID 32534455